CLINICAL TRIAL: NCT05344248
Title: A Randomized, Double Blinded, Multi-center, Placebo Controlled, Phase Ib/II Clinical Study to Evaluate the Safety, Tolerability, Efficacy and Pharmacokinetic Profiles of Multiple Doses of JS005 in Patients With Moderate to Severe Plaque Psoriasis
Brief Title: Safety, Tolerance, Efficacy and Pharmacokinetics of JS005 Multiple Dosing
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JS005-002-Ib/II
Record Dates: First submitted 2022-03-31; First posted 2022-04-25 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-03

CONDITIONS: Moderate to Severe Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JS005 (recombinant humanized monoclonal antibody against IL-17A) (Experimental): Ib：60mg、150mg、300mg、600mg；Each patient can only receive multiple doses at one dose level.Each patient received weekly dosing (QW) at weeks 0, 1, 2, 3, and 4, and quad-weekly dosing (Q4W) beginning at week 5 through week 12。 II：Multiple subcutaneous injections of the study drug and placebo in two doses of 300mg and 150mg were performed.Each patient can only receive multiple doses at one dose level.Weekly dosing (QW) was given at 0, 1, 2, 3, and 4 weeks, and quad-weekly dosing (Q4W) was given from 5 weeks to 12 weeks.
  Interventions: Biological: JS005 (recombinant humanized monoclonal antibody against IL-17A)
- Placebo (Placebo Comparator): Ib：60mg、150mg、300mg、600mg；Each patient can only receive multiple doses at one dose level.Each patient received weekly dosing (QW) at weeks 0, 1, 2, 3, and 4, and quad-weekly dosing (Q4W) beginning at week 5 through week 12。 II：Multiple subcutaneous injections of the study drug and placebo in two doses of 300mg and 150mg were performed.Each patient can only receive multiple doses at one dose level.Weekly dosing (QW) was given at 0, 1, 2, 3, and 4 weeks, and quad-weekly dosing (Q4W) was given from 5 weeks to 12 weeks.
  Interventions: Biological: JS005 placebo

INTERVENTIONS:
Biological: JS005 (recombinant humanized monoclonal antibody against IL-17A) — Subcutaneous injection
  Arms: JS005 (recombinant humanized monoclonal antibody against IL-17A)
Biological: JS005 placebo — Subcutaneous injection
  Arms: Placebo

SUMMARY:
JS005-002 is a randomized, double-blinded, placebo-controlled phase Ib/II clinical study to evaluate the safety, tolerability, efficacy and pharmacokinetic profiles of multiple doses of JS005 (recombinant humanized anti-IL-17A monoclonal antibody) Injection in patients with moderate to severe psoriasis.

DETAILED DESCRIPTION:
This study includes a total of two parts, the first part is a double-blinded, placebo-controlled, multi-dose escalation study to evaluate the safety, preliminary efficacy and pharmacokinetic profiles after multiple doses in patients with moderate to severe psoriasis; the second part is a randomized, double-blinded, controlled study, with proposed high-, middle- and low-dose groups and placebo group based on the clinical effective dose determined in the first part, to evaluate the efficacy and safety of multiple doses of test drug in patients with moderate to severe psoriasis.

Part I of study (phase Ib):

A total of 4 dose groups are pre-specified in Part I of this study, i.e., 60 mg, 150 mg, 300 mg and 600 mg; multiple doses will be administered subcutaneously on abdomen. A total of 40 patients are planned to be enrolled, including 6 and 2 patients receiving test drug and placebo in 60 mg and 600 mg dose groups, respectively, 9 and 3 patients receiving test drug and placebo in the other two dose groups, respectively. Each patient can receive multiple doses at only one dose level.

Part II of study (phase II):

Based on the safety data of phase Ib study and the efficacy analysis of ER modeling, 300mg and 150mg of the test drug will be selected. A multi-center, double-blind, placebo-controlled phase II study was conducted. The patients will be radomized in a 1:1:1 ratio to receive 300mg, 150mg doses of the study drug or placebo. A total of 126 patients will be enrolled in phase II study, with 42 patients in each group. 300mg, 150mg doses of the study drug or placebo will be administered abdominal subcutaneously with multiple dosing. Each patient can receive multiple doses at only one dose level.

ELIGIBILITY:
Inclusion criteria:

1. Male and female patients aged 18 ~ 75 years (inclusive, age limited to 18 ~ 60 years in Part I of the study);
2. Body mass index (BMI) = weight (kg)/ height 2 (m2), ranging from 18~30 kg/m2 (inclusive) at screening;
3. Being able to understand the content of the study and voluntary to sign the informed consent form; meanwhile, being able to complete the study as required in the protocol;
4. Having been diagnosed as chronic plaque psoriasis for at least 6 months prior to screening;
5. Being eligible for systemic therapy. Defined as moderate to severe chronic plaque psoriasis poorly controlled with local therapy and/or phototherapy and/or previous systemic therapy;
6. At screening, moderate to severe plaque psoriasis will be defined as followings: PASI score ≥ 12, PGA score ≥ 3 (in accordance with 0 ~ 5-point scale), and body surface area (BSA) affected by plaque psoriasis ≥10%;
7. No plan of pregnancy and being willing to use effective contraceptive measures for patients (including partners) from signature of informed consent to 6 months after administration of investigational product, see Appendix 7 for the specific contraceptive measures.

Exclusion criteria:

1. Prior biologic therapy (Secukinumab or Ixekizumab) that directly targets il-17 monoclonal antibody or IL-17 receptor at any time;
2. Use of a therapeutic biologic within 12 weeks prior to screening, or random administration of the drug during the elimination phase (5 half-lives), whichever is longer;
3. Participated in any other clinical study with investigational drug intervention within 12 weeks prior to screening, or the investigational drug was in the elimination phase (5 half-lives) at the time of randomization, whichever is longer;
4. Have received live vaccine within 12 weeks prior to screening, or plan to receive live vaccine within 12 weeks after administration of the last experimental drug;
5. Any infection requiring hospitalization, antiviral or antibiotic treatment within 30 days prior to screening (such as pneumonia, cellulitis, bone and joint infection, etc., and the investigator determined that the patient had low immune function and participation in this study might lead to unacceptable risks);
6. Received systemic treatment of Chinese herbal medicine for psoriasis within 30 days or external medication for psoriasis within 14 days prior to screening;
7. Have received systemic treatment for psoriasis within 30 days prior to screening or were using a prohibited treatment at the time of screening.As UV exposure is one of the contraindication treatments, patients who do not wish to limit their UV exposure (e.g., sunbathing and/or using tanning devices) during the study period will be excluded;
8. Non-chronic plaque psoriasis (e.g. Pustular psoriasis, erythrodermic psoriasis and intravenous psoriasis) at the time of screening;
9. Drug psoriasis (new or aggravated psoriasis caused by beta blockers, calcium channel inhibitors or lithium) at the time of screening;
10. The presence of other skin problems (e.g. skin infection, seborrheic dermatitis, severe allergic skin disease, etc.) that may interfere with the evaluation of psoriasis;
11. A history of inflammatory bowel disease, Crohn's disease, or other persistent active autoimmune disease;
12. Have a history of Tubercle bacillus (TB) infection, or chest imaging examination suggested TB infection during screening, or tuberculosis screening suggested latent tuberculosis infection;
13. History of transplantation of vital organs (such as heart, lung, liver, kidney, etc.);
14. A history or symptoms of malignancy in any organ system at the time of screening, whether or not it has been treated within the past 5 years, and whether or not there are signs of local recurrence or metastasis;
15. Having other significant medical problems at the time of screening, including, but not limited to, uncontrolled hypertension (systolic blood pressure ≥160mmHg and/or diastolic blood pressure ≥95mmHg), congestive heart failure (New York heart association status class III or IV);
16. Medical history and past history suggest other major diseases, including but not limited to gastrointestinal, renal, liver, neurological, hematological, endocrine, pulmonary, immune, psychiatric or cardiovascular and cerebrovascular diseases. The researcher considers that participation in this study would pose unacceptable risks to patients or significantly affect the study results;
17. Has undergone any major surgery within 8 weeks prior to screening, or is required to undergo such surgery during the study period, which the investigator and sponsor have confirmed may pose unacceptable risks to the patients;
18. Patients with serum creatinine above the upper limit of normal at screening time.Platelet & LT during screening;100 x109/L, neutrophils <1.5x109 /L, or hemoglobin <85g/L, ALT or AST level increased ≥ 2 times the upper limit of normal value;
19. Abnormal electrocardiogram during screening was considered clinically significant by the investigator, and participation in the study may bring unacceptable risks to the patients;
20. At the time of screening, HBV DNA copy number was detected in persons who were positive for human immunodeficiency virus antibody (ANTI-HIV), hepatitis C virus antibody (anti-HCV), hepatitis B surface antigen (HBsAg) or HBcAb (upper limit of reference value of each hospital for quantitative test line);
21. Known to suffer from moderate to severe allergic diseases or hypersensitivity reactions;
22. Known history of allergy or hypersensitivity to study drugs, other monoclonal antibodies and therapeutic protein preparations (human serum albumin, cytokines, interleukins, etc.);
23. Screening and randomization of female patients with β -human Chorionic Gonadotropin (β-HCG) positivity or breastfeeding;
24. Blood loss or blood donation within the last 3 months & GT;400mL, or patients who had received blood transfusion, or who planned to donate blood during the study;
25. Any other conditions considered unsuitable for study participation by the investigator, such as patients with other potential compliance problems, inability to complete all examinations and evaluations as required by the protocol, or uncontrolled neuropsychiatric or psychological disorders, present uncontrollable risks of study participation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2022-10-28 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
the numbers of adverse event(AE) | 0-24 weeks
  Safety evaluation will be documented as numbers of adverse event(AE)
II: The proportion of patients with at least PASI 75 at Week 12 | From week 0 to week 12
  The Proportion of patients with at least 75% improvement in PASI (PASI 75) at Week 12

SECONDARY OUTCOMES:
Ib: PK evaluation: Cmax | 0-24 weeks
  Maximum Plasma Concentration (Cmax)
Ib: PD evaluation: level of IL-17A | 0-24 weeks
  Population pharmacokinetic parameters will be provided and individual pharmacokinetic reports will be provided
Ib: PASI score response criteria | 0-24 weeks
  Mean change in PASI score from baseline at Week 12, 16 and 24.
Ib: Proportion of Patients achieving PASI 75 | 0-24 weeks
  Proportion of patients achieving PASI 75 at Week 12, 16 and 24.
Ib: Proportion of Patients achieving PASI 90/100 | 0-24 weeks
  Proportion of patients achieving PASI 90/100 at Week 12, 16 and 24.
Ib: Proportion of patients with PGA score | 0-12 weeks
  Proportion of patients with PGA score of 0 or 1 at Week 12
Ib: Mean change from baseline in body surface area (BSA) | 0-24 weeks
  Mean change from baseline in body surface area (BSA) affected by psoriasis at Week 12, 16 and 24
Ib: Proportion of patients with DLQI score | 0-24 weeks
  Proportion of patients with DLQI score of 0 or 1 at Week 12, 16 and 24
Ib: Time to ADA occurrence after drug administration | 0-24 weeks
  Time to ADA occurrence after drug administration.
Ib: Time to Nab occurrence after drug administration. | 0-24 weeks
  Time to Nab occurrence after drug administration.
II: Proportion of Patients achieving PASI 90 | 0-20 weeks
  Proportion of PASI 90 patients at week 12, 16, and 20
II: Proportion of patients with PGA score | 0-20 weeks
  Proportion of patients with PGA score of 0 or 1 at Week 12, 16 and 20
II: Patients achieving PASI 75 | 0-20 weeks
  Proportion of patients achieving PASI 75 at Week 16 and 20.
II: PASI score response criteria | 0-20 weeks
  Mean change in PASI score from baseline at Week 12, 16 and 20.
II: PASI and/or with PGA score response criteria | 0-20 weeks
  Proportion of patients meeting PASI75/90/100 and/or with PGA score of 0 or 1 at Week 12, 16 and 20
II: BSA response criteria | 0-20 weeks
  Change in BSA from baseline at Week 12, 16 and 20
Proportion of patients with DLQI score | 0-20 weeks
  Proportion of patients with DLQI score of 0 or 1 at Week 12, 16 and 20
II: The numbers of adverse event(AE). | 0-20 weeks
  Safety evaluation will be documented as numbers of adverse event(AE).
II: PK evaluation: Cmax | 0-20 weeks
  Maximum Plasma Concentration (Cmax)
II: PD evaluation: IL-17A | 0-20 weeks
  Population pharmacokinetic parameters will be provided and individual pharmacokinetic reports will be provided
II: Time to ADA occurrence after drug administration. | 0-20 weeks
  Time to ADA occurrence after drug administration.
Ib:PK evaluation: AUC0-inf | 0-24 weeks
  Area under the plasma concentration versus time curve (AUC0-inf)
Ib: Percentage of patients with positive ADA after drug administration. | 0-24 weeks
  Analysis of anti-drug antibody (ADA)
Ib: Percentage of patients with positive Nab after drug administration. | 0-24 weeks
  Detection of neutralizing antibody (Nab)
II: PK evaluation: AUC0-inf | 0-20 weeks
  Area under the plasma concentration versus time curve (AUC0-inf)
II: Percentage of patients with positive ADA after drug administration. | 0-20 weeks
  Analysis of anti-drug antibody (ADA)

CONTACTS AND LOCATIONS:
Locations (22):
- China (22):
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Beijing Tsinghua Changgung Hospita, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Dermatology Hospital of Southern Medical University, Guangzhou, Guangdong
  - The First Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Second Affiliated Hospital of Harbin Medical University, Haerbin, Heilongjiang
  - Dermatology Hospital, Chinese Academy of Medical Sciences, Nanjing, Jiangsu
  - Affiliated Hospital of Jiangsu University, Zhenjiang, Jiangsu
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - First Hospital of Jilin University, Changchun, Jilin
  - Dermatology Hospital affiliated to Shandong First Medical University, Jinan, Shandong
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai Skin Disease Hospital, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - Affiliated Hospital of Tianjin Academy of Traditional Chinese Medicine, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang